CLINICAL TRIAL: NCT01819649
Title: Prevention of Cancer by Intervention With Selenium - A Pilot Study in a Danish Population
Brief Title: Selenium in the Prevention of Cancer
Acronym: DK PRECISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Danish Cancer Society (Other); University of Southern Denmark (Other); K. A. Rohde's and wife's Foundation (Other); The County of Funen, Denmark (Other Government); Cypress Systems, USA (Unknown); The Dagmar Marshall Foundation (Other); The N. O. Andersen Foundation (Unknown); The Danish Directory of Food and Agriculture (Unknown); The Foundation of Clinical Experimental Cancer Research, Odense (Unknown); The Foundation of Lily Benthine Lund (Unknown); The Memory Foundation of Merchant Brogaard (Unknown); Pharma Nord (Industry)
Responsible Party: Principal Investigator, Søren Cold, M.D. PhD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OUH-DK-PILOT-PRECISE
Record Dates: First submitted 2013-01-23; First posted 2013-03-27 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Cancer
Keywords: selenium; selenium supplementation; randomised controlled trial; prevention
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: AMENDMENT TO STUDY DESIGN: Towards the end of the intervention period, it was decided to follow-up participants for an additional ten years via Danish public registries for data on morbidity and mortality.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Selenium enriched-yeast tablet; SelenoPRECISE 100 mcg/d (Experimental)
  Interventions: Dietary Supplement: SelenoPRECISE selenium-enriched yeast tablet, Pharma Nord Denmark A/S
- Selenium enriched-yeast tablet; SelenoPRECISE 200 mcg/d (Experimental)
  Interventions: Dietary Supplement: SelenoPRECISE selenium-enriched yeast tablet, Pharma Nord Denmark A/S
- Selenium enriched-yeast tablet; SelenoPRECISE 300 mcg/d (Experimental)
  Interventions: Dietary Supplement: SelenoPRECISE selenium-enriched yeast tablet, Pharma Nord Denmark A/S
- Yeast tablet (Placebo Comparator)
  Interventions: Dietary Supplement: SelenoPRECISE selenium-enriched yeast tablet, Pharma Nord Denmark A/S

INTERVENTIONS:
Dietary Supplement: SelenoPRECISE selenium-enriched yeast tablet, Pharma Nord Denmark A/S

SUMMARY:
This is a pilot study proceeding an intended international trial.

Hypothesis: Daily intake of selenium supplementation in the form of selenium-enriched yeast tablets will reduce the risk of cancer in healthy individuals.

Objective: The objective of this pilot study was to assess the viability of a full scale randomised trial.

AMENDMENT TO STUDY OBJECTIVE: Mortality analysis during intervention and follow-up as specified in the sections concerning study design and outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* WHO performance status 0 or 1
* No active liver- or kidney disease (Serum ALAT (alanine aminotransferase), alkalic phosphatase, bilirubin, creatinin or urea within 2 S.D of laboratory reference range)
* No previous cancer diagnosis
* No known HIV-infection
* Participant must understand oral and written information
* Participant must not use selenium supplementation of above 50 mcg/d
* Participant must give written consent prior to inclusion

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 1998-11; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Viability of full scale study | At five years intervention
  At five years intervention (last participant last visit was june 2004) viability of full scale study was assessed according to the drop out rate, cost etc. of this pilot study.

SECONDARY OUTCOMES:
AMENDMENT TO OUTCOME MEASURES: Mortality analysis. | Up to 17 years
  Study participants will be followed up for mortality from the date of randomization in 1998-1999 through March 31, 2015. Vital status and date of death will be obtained from the Danish Civil Registration System. Information on the underlying cause of death will be obtained from the Danish Registry of Causes of Death through December 31, 2010 and from participant medical charts from January 1, 2011. Cause of death will be classified according to the 10th Revision of the International Classification of Diseases as death due to cancer (codes C00-C97), CVD (I00-I99), and all other causes.

CONTACTS AND LOCATIONS:
Locations (1):
- Selenium Centre, Odense University Hospital, Odense C, Denmark

REFERENCES:
- [Derived] Cold F, Winther KH, Pastor-Barriuso R, Rayman MP, Guallar E, Nybo M, Griffin BA, Stranges S, Cold S. Randomised controlled trial of the effect of long-term selenium supplementation on plasma cholesterol in an elderly Danish population. Br J Nutr. 2015 Dec 14;114(11):1807-18. doi: 10.1017/S0007114515003499. Epub 2015 Sep 30. PMID 26420334